CLINICAL TRIAL: NCT01239420
Title: Norwegian Cardio-Respiratory Arrest Study (NORCAST)
Brief Title: Norwegian Cardio-Respiratory Arrest Study
Acronym: NORCAST
Status: Active, not recruiting | Type: Observational
Sponsor: Oslo University Hospital (Other)
Responsible Party: Principal Investigator, Espen Rostrup Nakstad, MD, Oslo University Hospital
Other Study IDs: REK S-O A Ref 2010/1116a
Record Dates: First submitted 2010-11-10; First posted 2010-11-11 (Estimated); Last update posted 2024-04-05 (Actual); Status verified 2024-04

CONDITIONS: Cardiac Arrest; Respiratory Arrest; Coma
MeSH Terms: conditions — Heart Arrest; Apnea; Coma

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Serum, plasma, blood (PaxGene). For future identification of biochemical markers in prognostication after cardiorespiratory arrest. For future identification of biochemical markers for cardiac arrest (primarily serum, but also on mRNA-level).
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of this study is to evaluate the use of combined clinical-neurological, neurophysiologic, neuroradiological and biochemical markers in prognostication after cardio- and/or respiratory arrest.

DETAILED DESCRIPTION:
Cardiac arrest (CA) is a leading cause of death, affecting about 700.000 individuals each year in Europe. Acute Myocardial Infarction (AMI) and primary arrhythmia are the most common causes of CA, whereas respiratory arrest is a leading cause of secondary CA. Patients who have undergone cardiopulmonary resuscitation (CPR) often remain unconscious after hospital admission, either as a result of severe permanent brain damage or a merely reversible metabolic disturbance due to post-ischemic global reperfusion. Early prediction of neurological and cardiac outcome remains a difficult task for physicians. The decision to continue, limit or terminate intensive care therapy carries huge ethical and socioeconomic implications. Optimal emergency cardiovascular care, cardiac failure therapy and CA prevention after hospitalisation also remain difficult issues for cardiologists and intensive care doctors.

In this prospective study running from 2010, both prognostication and in-hospital treatment are studied in a population of 261 patients with out-of-hospital cardio-respiratory arrest. The use of combined clinical-neurological, neurophysiologic, neuroradiological and biochemical markers is studied to asses whether a poor neurological outcome (Cerebral Performance Category 3-5) can be predicted with ~100% specificity and a sensitivity that is sufficient for practical clinical use.

Pre-disposing and triggering causes of cardiorespiratory arrest are also registered. Patients with pre-existing conditions coherent with prophylactic ICD implementation under current international guidelines will be identified, in order to assess and further improve ICD-prophylactic treatment in Norway. The potential benefit of invasive PICCO-monitoring after CA will also be evaluated, and a subproject identifying biomarkers for CA risk has been established. NIRS (Near-Infrared spectroscopy) will also be used to register cerebral oxygenation in the early days after cardiorespiratory arrest.

The overall aim of the NORCAST study is to provide physicians with better tools to asses cardiac and neurological outcome as early and as accurate as possible.

All alive study patients are invited to long-term follow-up consultaions after 6 months, after 4 years, and after 10 years. The consultations will include study examinations, structured interviews and questionnaires. Questionnaires will also be used for next of kin.

ELIGIBILITY:
Inclusion Criteria:

* prehospital cardial resuscitation
* prehospital pulmonary resuscitation
* ROSC before/on admission to hospital
* > 18 years of age

Exclusion Criteria:

* death on admission to hospital
* arrhythmic cardiac arrest with ALS < 5min and spontaneous awakening
* in-hospital cardiac arrest
* trauma patients

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients admitted after pre-hospital cardio/respiratory arrest.
Sampling Method: Probability Sample
Enrollment: 261 (Actual)
Dates: Start 2010-09; Primary Completion 2018-08 (Actual); Study Completion 2028-12 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Dag Jacobsen, MD, PhD, Study Director — Oslo University Hospital - Ulleval, Norway; Kjetil Sunde, MD, PhD, Study Director — Oslo University Hospital - Ulleval, Norway
Locations (1):
- Oslo University Hospital - Ulleval, Oslo, Norway

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Beitland S, Nakstad ER, Berg JP, Troseid AS, Brusletto BS, Brunborg C, Lundqvist C, Sunde K. Urine beta-2-Microglobulin, Osteopontin, and Trefoil Factor 3 May Early Predict Acute Kidney Injury and Outcome after Cardiac Arrest. Crit Care Res Pract. 2019 May 7;2019:4384796. doi: 10.1155/2019/4384796. eCollection 2019. PMID 31205786
- [Derived] Beitland S, Waldum-Grevbo BE, Nakstad ER, Berg JP, Troseid AS, Brusletto BS, Brunborg C, Andersen GO, Sunde K. Urine biomarkers give early prediction of acute kidney injury and outcome after out-of-hospital cardiac arrest. Crit Care. 2016 Oct 5;20(1):314. doi: 10.1186/s13054-016-1503-2. PMID 27716377
- [Derived] Staer-Jensen H, Nakstad ER, Fossum E, Mangschau A, Eritsland J, Draegni T, Jacobsen D, Sunde K, Andersen GO. Post-Resuscitation ECG for Selection of Patients for Immediate Coronary Angiography in Out-of-Hospital Cardiac Arrest. Circ Cardiovasc Interv. 2015 Oct;8(10):e002784. doi: 10.1161/CIRCINTERVENTIONS.115.002784. PMID 26453688